CLINICAL TRIAL: NCT03315312
Title: FISSURE-Project. Improved Dental Decay Management in Dental Service for Children: Fissure Sealants or Fluoride Varnish?
Brief Title: Occlusal Caries Management in First Permanent Molars in Child Dental Care
Acronym: FISSURE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oral Health Centre of Expertise in Eastern Norway (Other)
Collaborators: Public Dental Service, Hedmark (Unknown); Public Dental Service, Oppland (Unknown); Public Dental Service, Østfold (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FISSURE
Record Dates: First submitted 2017-10-11; First posted 2017-10-20 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Dental Caries Pit and Fissure; Dental Caries in Children
MeSH Terms: interventions — Fluorides, Topical; Pit and Fissure Sealants

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fissure sealant (Active Comparator)
  Interventions: Drug: Fissure Sealants
- Fluoride varnish (Experimental)
  Interventions: Drug: Fluoride Varnishes

INTERVENTIONS:
Drug: Fluoride Varnishes — Fluoride varnish is randomly applied on randomly selected first permanent molar. This study uses a natural clinical setting, where clinicians use methods and procedures that are routinely applied in public dental clinics.
  Arms: Fluoride varnish
Drug: Fissure Sealants — Resin-based fissure sealant is applied on contra-lateral first permanent molar and each child serves as its own control. This study uses a natural clinical setting, where clinicians use methods and procedures that are routinely applied in public dental clinics.
  Arms: Fissure sealant

SUMMARY:
Occlusal caries management in first permanent molars: a pragmatic randomized clinical trial in child dental care

Aim of the present study is to evaluate the effectiveness of fissure sealants and fluoride varnish in a pragmatic randomized clinical trial and evaluate whether some specific patient groups benefit more from any particular treatment.

The high risk children (having a previous caries experience at 5 years of age) from 2009, 2010 and 2011 birth cohorts (6-, 7- and 8-year-olds) from three counties (Østfold, Oppland and Hedmark) are selected. Children with at least two erupted first permanent molars in the same jaw randomly receive resin-based sealant or a fluoride varnish (Duraphat) during a routine dental examination. Children who already developed caries, had restorations or fissure sealants placed in first molars were excluded from the present study.

Fluoride varnish and resin-based fissure sealants are randomly applied on contra-lateral teeth where each child serves as its own control. This study uses a natural clinical setting, where clinicians use methods and procedures that are routinely applied in public dental clinics. The study is approved by the Regional Committee for Medical Research Ethics South East (2016/2002/REK sør-øst C).

Sample size calculations: Based on the assumption that 80% of the treated teeth do not get caries and that 10% difference in caries development constitutes a clinically meaningful difference, it is required to recruit 180 participants in the study for the split-mouth design. Considering a potential maximum of annual 20% drop-out rate and a 3-years follow-up, the study will need to recruit 400 participants in order to have at least 206 children at the 3 years of follow-up.

Treatments are provided by either dentists or dental hygienists during routine dental examinations. Caregivers of eligible children are informed about the study, the participation is voluntary and an informed written parental consent is obtained in accordance with the directions of the Regional Committee for Medical Research Ethics. In this study, a clinician selects a random treatment for the first tooth by choosing one of the two cards, while a collateral tooth receives an alternative treatment. Subsequently, treatments provided and materials used are recorded on a treatment registration form. During this study, clinicians follow their conventional clinical procedures for applying sealants or fluoride varnish. Information on patient's caries experience and quality of oral hygiene are recorded on treatment registration form. Fluoride varnish is applied three times, at baseline, 6 months and 12 months.

Caries on occlusal surfaces of first molars detected at later 24 and 36 months follow-ups will be recorded in the follow-up registration form. The main study outcome is caries occurrence on occlusal tooth surfaces.

ELIGIBILITY:
Inclusion Criteria:

* The high risk children (having a previous caries experience at 5 years of age) with at least two erupted first permanent molars

Exclusion Criteria:

* Children who already developed caries, had restorations or fissure sealants placed in first molars are excluded from the present study.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 410 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dental caries incidence on occlusal surfaces of first molars | 12 months after application
  Decayed, missing and filled surfaces (DMFS) increment
Dental caries incidence on occlusal surfaces of first molars | 24 months after application
  Decayed, missing and filled surfaces (DMFS) increment
Dental caries incidence on occlusal surfaces of first molars | 36 months after application
  Decayed, missing and filled surfaces (DMFS) increment

CONTACTS AND LOCATIONS:
Locations (1):
- Public Dental Service clinics at Østfold county, Sarpsborg, Norway

IPD SHARING:
Plan to Share IPD: No